CLINICAL TRIAL: NCT05247814
Title: Individual Patient Risk Profiles for Adverse Drug Reactions: Establishing a Consecutive Research Cohort in an Interdisciplinary Polypharmacy Consultation Service of a Geriatric University Outpatient Department
Brief Title: Individual Risk Profiles for Adverse Drug Reactions in Geriatric Patients
Status: Not yet recruiting | Type: Observational
Sponsor: RWTH Aachen University (Other)
Collaborators: B. Braun Foundation (Other)
Responsible Party: Principal Investigator, Julia Stingl, Univ.-Prof. Dr. med., RWTH Aachen University
Other Study IDs: 21-216
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Polypharmacy; Pharmacogenetics; Pharmacogenomic Testing; Drug-Related Side Effects and Adverse Reactions
Keywords: Geriatric Assessment; Medication Adherence; Aged; Aged, 80 and over; Medication therapy management; Pharmacists; Geriatricians; Clinical Pharmacology; Medication reconciliation; Hospital pharmacy services; Hospital outpatient clinics; nterdisciplinary Health Team
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — DNA will be isolated from patients' blood samples. Patients will then be genotyped for relevant pharmacogenes focusing on drug metabolizing enzymes CYP2D6, 2C9, and 2C19 and other genes of clinical relevance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients admitted to interdisciplinary polypharmacy consultation service: Patients admitted to the Interdisciplinary Polypharmacy Consultation Service of the Department of Geriatric's University Outpatient Clinic in cooperation with the Institute of Clinical Pharmacology
  Interventions: Genetic: Pharmacogenomic testing of a panel of important pharmacogenes to detect genetic variants and evaluate the association between genetically predicted and measured drug metabolism; Other: Adverse Drug Reaction detection; Other: Falls Efficacy Scale International (FES-I)

INTERVENTIONS:
Genetic: Pharmacogenomic testing of a panel of important pharmacogenes to detect genetic variants and evaluate the association between genetically predicted and measured drug metabolism — All planned interventions are explorative analyses of biological and genetic risk profiles that can contribute to patients' individual risk for adverse drug reactions, i.e. due to variability in drug metabolism
Other: Adverse Drug Reaction detection — During appointments in the university outpatient clinic, patients will undergo a comprehensive adverse drug reaction (ADR) assessment based on an ADR diary they were handed at enrolment
Other: Falls Efficacy Scale International (FES-I) — The FES-I wil be obtained to estimate fear of falling

SUMMARY:
This project will generate a prospective cohort of geriatric patients with polypharmacy which will be characterized for vulnerability profiles of adverse drug reactions.

DETAILED DESCRIPTION:
Adverse drug reactions are common in older patients and can lead to severe outcomes such as falls, hospitalizations and death. They are dose-dependent and may for example be caused by inappropriate dosing due to a reduced kidney function. Also, the use of potentially inappropriate medications in older patients can result in a negative benefit-/ risk-ratio. Additionally, drug metabolism in older patients is altered due to a variety of reasons and pharmacogenetic variants of drug metabolizing enzymes can lead to a more than 10-fold interinidividual variation of drug clearance. The risk of the individual patient to experience an adverse drug reactions is determined by many reasons. Therefore, this study aims to identify patient risk profiles with regard to pharmacogenetics, drug interactions, impaired functional and cognitive status and individual drug metabolism.

Participants for this study will be consecutively recruited from patients admitted to the Interdisciplinary Polypharmacy Consultation Service of the Department of Geriatric's University Outpatient Clinic in cooperation with the Institute of Clinical Pharmacology. Regardless of their participation in this study, patients in the outpatient clinic will perform several tests and questionnaires following the comprehensive geriatric assessment. The purpose of the cohort study is to document and evaluate routine health data collected in the outpatient clinic for polypharmacy in geriatric patients (laboratory tests as well as a comprehensive medication history with therapy recommendations issued by a subsequent pharmaceutical council for both the patients and the primary care physicians).

Procedures conducted specifically for this study are a long-term capture and detailed history of all suspected adverse drug reactions, examining the fear of falling (FES-I questionnaire) and blood sampling for exploratory pharmacogenomic analyses (on cohort level, not patient diagnostics).

Aim of the long-term cohort of geriatric patients with polypharmacy is to identify risk profiles for adverse drug reactions that are specific for the population of older individuals.

ELIGIBILITY:
Inclusion Criteria:

* 70 years or older
* Current drug therapy with three or more drugs
* Being a patient in the interdisciplinary polypharmacy consultation service of the geriatric university outpatient clinic
* Sufficient mobility (minimum: Wheelchair mobility)
* Written informed consent of the patient or the legal representative

Exclusion Criteria:

* No sufficient communication possible
* Patients classified as terminally ill by the medical staff
* Patients, that are incapable to give their informed consent and who do not have a legal representative

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted to the Interdisciplinary Polypharmacy Consultation Service of the Department of Geriatric's University Outpatient Clinic in cooperation with the Institute of Clinical Pharmacology
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2032-02 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
Identification of vulnerability profiles of adverse drug reactions | February 2022 - February 2032
  To investigate patient-specific risk profiles for adverse drug reactions, the focus of this study is on analizing patients' functional and cognitive status, pharmacogenetics, and individual metabolic capacity (phenotype/genotype relationship).

CONTACTS AND LOCATIONS:
Overall Officials: Julia C. Stingl, MD, ScD, Principal Investigator — Institute of Clinical Pharmacology, University Hospital RWTH Aachen

IPD SHARING:
Plan to Share IPD: Undecided